CLINICAL TRIAL: NCT00360490
Title: A Multicenter, Randomized, Open Label, Parallel Group, Active Control Study to Evaluate the Efficacy and Safety of LNG IUS (Mirena®) as Compared to Medroxyprogesterone Acetate During 6 Cycles of Treatment in Patients With Idiopathic Menorrhagia
Brief Title: Study in Women With Idiopathic Menorrhagia to Determine the Reduction in Menstrual Blood Loss (MBL) After Treatment With the Levonorgestrel-releasing Intrauterine System (IUS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91518; 309849 (Other: Bayer); NCT00360620 (obsolete NCT alias)
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-11

CONDITIONS: Menorrhagia
Keywords: Idiopathic Menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — Levonorgestrel; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levonorgestrel Intrauterine System (LNG IUS) 20µg per 24 hours (Experimental): Initial release rate of 20µg Levonorgestrel IUS (Mirena, BAY86-5028) per day for 6 cycles.
  Interventions: Drug: Levonorgestrel IUS (Mirena, BAY86-5028)
- Medroxyprogesterone acetate (MPA) (Active Comparator): Medroxyprogesterone acetate (MPA, Provera), oral, 10mg per tablet on 10 consecutive days of each cycle for 6 cycles.
  Interventions: Drug: Medroxyprogesterone acetate

INTERVENTIONS:
Drug: Levonorgestrel IUS (Mirena, BAY86-5028) — Initial release rate of 20µg Levonorgestrel IUS (Mirena, BAY86-5028) per day for 6 cycles.
  Arms: Levonorgestrel Intrauterine System (LNG IUS) 20µg per 24 hours
Drug: Medroxyprogesterone acetate — Medroxyprogesterone acetate (MPA, Provera), oral, 10mg per tablet on 10 consecutive days of each cycle for 6 cycles.
  Arms: Medroxyprogesterone acetate (MPA)

SUMMARY:
The purpose of this study is to determine whether the levonorgestrel-releasing intrauterine system is effective in decreasing menstrual blood loss.

DETAILED DESCRIPTION:
Acronyms in the Adverse Event Section:

* IUCD Intrauterine Contraceptive Device
* MedDRA Medical Dictionary for Regulatory Activities

This study has previously been posted by Berlex, Inc. and Schering AG, Germany. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc., Schering AG Germany has been renamed to Bayer HealthCare AG, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Women who have >/= 80 mL blood loss during their menstrual cycles and desire contraception

Exclusion Criteria:

* Post menopausal menstrual cycle < 21 days or > 35 days
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (51):
- United States (35):
  - Tucson, Arizona
  - Beverly Hills, California
  - Carmichael, California
  - San Diego, California
  - Santa Monica, California
  - Torrance, California
  - Littleton, Colorado
  - Boynton Beach, Florida
  - Jacksonville, Florida
  - West Palm Beach, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Newburgh, Indiana
  - South Bend, Indiana
  - Amite, Louisiana
  - Marrero, Louisiana
  - Boston, Massachusetts
  - Saginaw, Michigan
  - Chesterfield, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - LasVegas, Nevada
  - Moorestown, New Jersey
  - New Brunswick, New Jersey
  - Winston-Salem, North Carolina
  - Medford, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Clarksville, Tennessee
  - Houston, Texas
  - Burlington, Vermont
  - Norfolk, Virginia
  - Seattle, Washington
- Argentina (2):
  - Buenos Aires, Argentina
  - Buenos Aires, Buenos Aires
- Brazil (2):
  - Curitiba, Paraná
  - Campinas, São Paulo
- Canada (9):
  - Bathurst, New Brunswick
  - Ottawa, Ontario
  - Toronto, Ontario
  - Mirabel, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Shawinigan, Quebec
  - Regina, Saskatchewan
- Mexico (3):
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - México, State of Mexico

REFERENCES:
- [Result] Endrikat J, Vilos G, Muysers C, Fortier M, Solomayer E, Lukkari-Lax E. The levonorgestrel-releasing intrauterine system provides a reliable, long-term treatment option for women with idiopathic menorrhagia. Arch Gynecol Obstet. 2012 Jan;285(1):117-21. doi: 10.1007/s00404-011-1902-1. Epub 2011 Apr 8. PMID 21475963
- [Result] Kaunitz AM, Bissonnette F, Monteiro I, Lukkari-Lax E, DeSanctis Y, Jensen J. Levonorgestrel-releasing intrauterine system for heavy menstrual bleeding improves hemoglobin and ferritin levels. Contraception. 2012 Nov;86(5):452-7. doi: 10.1016/j.contraception.2012.07.018. Epub 2012 Sep 7. PMID 22959906
- [Result] Kaunitz AM, Bissonnette F, Monteiro I, Lukkari-Lax E, Muysers C, Jensen JT. Levonorgestrel-releasing intrauterine system or medroxyprogesterone for heavy menstrual bleeding: a randomized controlled trial. Obstet Gynecol. 2010 Sep;116(3):625-632. doi: 10.1097/AOG.0b013e3181ec622b. PMID 20733445

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 807 subjects screened; 165 subjects randomized to either Levonorgestrel Intrauterine System (LNG IUS) or Medroxyprogesterone acetate (MPA) for treatment of idiopathic menorrhagia; 145 subjects completed study.
Period: Overall Study
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Started | 82 | 83
Completed | 73 | 72
Not Completed | 9 | 11
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 0 | 4
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA) | Total
Number analyzed (Participants) | 82 | 83 | 165
Age Continuous [Mean (Full Range); unit: years] | 38.3 [26 to 50] | 39.3 [26 to 53] | 38.8 [26 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 83 | 165
  Male | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m²] — There is one participant [patient identifier (pid) =11407] missing in Levonorgestrel Intrauterine System group.
  kg/m² | 27.19 (3.903) | 27.36 (4.610) | 27.28 (4.263)

OUTCOME MEASURES:

1. Primary Outcome: The Change in Absolute Value From Baseline Menstrual Blood Loss (MBL) to the End-of-study MBL (Cycle 6)
Description: The MBL for each cycle included intermenstrual bleeding in addition to withdrawal bleeding. Baseline MBL was the composite MBL measured during each of the cycles during the Screening Phase. End-of-study MBL was measured during Cycle 6 of the Treatment Phase.
Time Frame: Baseline and up to 6 months
Population: Among of the 165 Full Analysis Set (FAS) subjects, a total of 160 subjects (79 for LNG IUS and 81 for MPA) were available for the analysis. One subject in LNG IUS, and two subjects in MPA group were not available due to the missing of diary data, and 2 subjects in LNG IUS group were not available due to the invalid baseline data.
Measure: Median (Full Range); unit: milliliter (mL)
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 79 | 81
milliliter (mL) | -128.78 [-393.6 to 1242.2] | -17.7 [-271.5 to 78.6]
Statistical Analysis 1: Comparison: Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours vs Medroxyprogesterone Acetate (MPA); The null hypothesis: the absolute change from Baseline MBL to End of Study MBL is equal in the LNG IUS group and the MPA group; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Percentage of Patients With Successful Treatment
Description: End-of-study MBL < 80 mL and a decrease to a value no greater than 50% of the Baseline MBL was considered to be treatment success.
Time Frame: At 6 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 79 | 81
Percentage of participants | 84.8 | 22.2
Statistical Analysis 1: Comparison: Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours vs Medroxyprogesterone Acetate (MPA); The null hypothesis: the proportion of subjects with successful treatment is equal in the LNG IUS group and the MPA group; Test type: Superiority or Other; p < 0.001, Chi-squared; Risk Difference (RD) = 62.59, 95% CI [50.56 to 74.61]

3. Secondary Outcome: Percent Change From Baseline MBL to End of Study MBL (Cycle 6)
Description: The percent change = {(End of Study MBL - Baseline MBL)/Baseline MBL} x 100.
Time Frame: Baseline and up to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 79 | 81
Percent change | -70.75 (88.31) | -21.54 (35.79)
Statistical Analysis 1: Comparison: Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours vs Medroxyprogesterone Acetate (MPA); The null hypothesis: the percent change from Baseline MBL to End of Study MBL is equal in the LNG IUS group and the MPA group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -49.2, 95% CI [-70.2 to -28.3]

4. Secondary Outcome: Absolute Change From Baseline MBL to Mid-study MBL (Cycle 3)
Description: The MBL for each cycle included intermenstrual bleeding in addition to withdrawal bleeding. Mid-study MBL was measured during Cycle 3 of the Treatment Phase.
Time Frame: Baseline and up to 3 months
Population: as for outcome 1
Measure: Median (Full Range); unit: milliliter (mL)
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 79 | 81
milliliter (mL) | -115.13 [-405.8 to 54.4] | -3.15 [-270.9 to 146.7]
Statistical Analysis 1: Comparison: Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours vs Medroxyprogesterone Acetate (MPA); The null hypothesis: the absolute change from Baseline MBL to Mid-study MBL is equal in the LNG IUS group and the MPA group; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percent Change From Baseline MBL to Mid-study MBL (Cycle 3)
Description: The percent change = {(Mid-study MBL - Baseline MBL)/Baseline MBL} x 100.
Time Frame: Baseline and up to 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 79 | 81
Percent change | -61.71 (41.76) | -11.11 (42.46)
Statistical Analysis 1: Comparison: Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours vs Medroxyprogesterone Acetate (MPA); The null hypothesis: the percent change from Baseline MBL to Mid-study MBL is equal in the LNG IUS group and the MPA group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -50.6, 95% CI [-63.8 to -37.4]

6. Secondary Outcome: Percentage of Subjects Who Completed the Study in Levonorgestrel Intrauterine System (LNG IUS) Group
Time Frame: Baseline and up to 6 months
Population: Among of the 165 Full Analysis Set (FAS) subjects, a total of 160 subjects (79 for LNG IUS and 81 for MPA) were available for the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours
Number analyzed (Participants) | 79
percentage of participants
  0 days | 97.53
  30 days | 95.06
  60 days | 93.83
  90 days | 92.59
  120 days | 91.36
  150 days | 90.12
  180 days | 90.12

7. Secondary Outcome: Total Number of Bleeding Days
Description: In the LNG IUS group, each cycle has 30 days. In the MPA group, each menstrual cycle starts on the 1st bleeding day (withdrawal bleeding) and lasts until the last non-bleeding day before next withdrawal bleeding starts.
Time Frame: Baseline and up to 6 months
Population: Among of the 165 Full Analysis Set (FAS) subjects, a total of 163 subjects (81 for LNG IUS and 82 for MPA) were available for the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 81 | 82
days
  Baseline | 5.64 (1.573) | 5.64 (1.280)
  Cycle 1 | 10.23 (5.784) | 5.17 (1.349)
  Cycle 2 | 7.88 (5.256) | 5.15 (1.459)
  Cycle 3 | 5.92 (4.505) | 5.25 (1.648)
  Cycle 4 | 4.77 (4.455) | 4.82 (1.591)
  Cycle 5 | 3.77 (4.560) | 4.89 (1.325)
  Cycle 6 | 4.16 (4.631) | 5.29 (1.835)

8. Secondary Outcome: Total Number of Spotting and Bleeding Days
Description: as for outcome 7
Time Frame: Baseline and up to 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 81 | 82
days
  Baseline | 6.30 (1.744) | 6.80 (1.990)
  Cycle 1 | 19.70 (7.894) | 6.65 (2.265)
  Cycle 2 | 17.46 (7.293) | 7.46 (2.294)
  Cycle 3 | 11.89 (7.415) | 6.92 (2.569)
  Cycle 4 | 10.42 (6.426) | 6.66 (2.372)
  Cycle 5 | 10.25 (7.359) | 6.89 (2.482)
  Cycle 6 | 8.58 (7.024) | 6.90 (2.834)

9. Secondary Outcome: Total Number of Spotting Days
Description: as for outcome 7
Time Frame: Baseline and up to 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 81 | 82
days
  Baseline | 1.23 (1.191) | 1.84 (1.638)
  Cycle 1 | 9.47 (6.933) | 1.48 (1.613)
  Cycle 2 | 9.58 (7.073) | 2.31 (2.004)
  Cycle 3 | 7.27 (6.421) | 2.27 (2.150)
  Cycle 4 | 5.65 (5.079) | 1.84 (1.767)
  Cycle 5 | 6.48 (5.869) | 2.00 (2.297)
  Cycle 6 | 5.38 (6.330) | 2.23 (2.532)

10. Secondary Outcome: Total Number of Bleeding Episodes
Description: A bleeding episode is defined as a light, normal or heavy bleeding, during a minimum of one day. In the LNG IUS group, each cycle has 30 days. In the MPA group, each menstrual cycle starts on the 1st bleeding day (withdrawal bleeding) and lasts until the last non-bleeding day before next withdrawal bleeding starts.
Time Frame: Baseline and up to 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: number of bleeding episodes
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 81 | 82
number of bleeding episodes
  Baseline | 1.01 (0.075) | 1.03 (0.115)
  Cycle 1 | 1.75 (0.707) | 0.98 (0.222)
  Cycle 2 | 0.88 (0.653) | 1.01 (0.194)
  Cycle 3 | 0.99 (0.647) | 0.97 (0.228)
  Cycle 4 | 0.76 (0.615) | 0.99 (0.202)
  Cycle 5 | 0.77 (0.755) | 1.01 (0.208)
  Cycle 6 | 0.70 (0.739) | 1.04 (0.359)

11. Secondary Outcome: Percent Change in Hemoglobin
Time Frame: Baseline and up to 6 months
Population: Among of the 165 Full Analysis Set (FAS) subjects, a total of 150 subjects (75 for LNG IUS and 75 for MPA) were available for the analysis.
Measure: Median (Full Range); unit: percent change
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 75 | 75
percent change
  Baseline to cycle 3 | 3.82 [-7.1 to 25.3] | 1.65 [-15.4 to 20.2]
  Cycle 3 to cycle 6 | 3.28 [-7.9 to 18.0] | 0.83 [-11.0 to 16.9]
  Baseline to cycle 6 | 7.50 [-3.6 to 44.0] | 1.87 [-17.9 to 33.3]

12. Secondary Outcome: Percent Change in Hematocrit
Time Frame: Baseline and up to 6 months
Population: as for outcome 11
Measure: Median (Full Range); unit: percent change
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 75 | 75
percent change
  Baseline to cycle 3 | 4.9 [-8 to 21] | 0.0 [-15 to 21]
  Cycle 3 to cycle 6 | 2.4 [-11 to 13] | 0.0 [-14 to 18]
  Baseline to cycle 6 | 5.4 [-7 to 26] | 0.0 [-21 to 26]

13. Secondary Outcome: Percent Change in Serum Ferritin
Time Frame: Baseline and up to 6 months
Population: Among of the 165 Full Analysis Set (FAS) subjects, a total of 148 subjects (75 for LNG IUS and 73 for MPA) were available for the analysis.
Measure: Median (Full Range); unit: percent change
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 75 | 73
percent change
  Baseline to cycle 3 | 13.8 [-67 to 300] | 0.0 [-78 to 380]
  Cycle 3 to cycle 6 | 48.3 [-51 to 293] | 16.7 [-78 to 560]
  Baseline to cycle 6 | 68.8 [-52 to 1440] | 14.3 [-87 to 540]

14. Secondary Outcome: Percentage of Patients With Improvement in the Investigator Global Assessment Scale
Description: "Improved" is classified as 'very much improved', 'much improved', or 'improved' and "not improved" is classified as 'no change', 'worse', 'much worse', or 'very much worse'
Time Frame: Up to 6 months
Population: Among of the 165 Full Analysis Set (FAS) subjects, a total of 160 subjects (78 for LNG IUS and 82 for MPA) were available for the analysis.
Measure: Number; unit: percentage
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 78 | 82
percentage
  Cycle 3 | 94.7 | 71.2
  Cycle 6 | 93.6 | 61.0

15. Secondary Outcome: Percentage of Patients With Improvement in the Patients Overall Assessment Scale
Description: as for outcome 14
Time Frame: Up to 6 months
Population: as for outcome 14
Measure: Number; unit: percentage
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Number analyzed (Participants) | 78 | 82
percentage
  Cycle 3 | 93.3 | 74.0
  Cycle 6 | 93.6 | 67.1
Statistical Analysis 1: Comparison: Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours vs Medroxyprogesterone Acetate (MPA); A two-sided 95% confidence interval for the improvement rate will be provided for cycle 6; Test type: Superiority or Other; Risk Difference (RD) = 26.06, 95% CI [14.75 to 37.36]

ADVERSE EVENTS:
Arm/Group | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours | Medroxyprogesterone Acetate (MPA)
Serious Adverse Events (participants affected / at risk) | 1/82 | 0/83
Other Adverse Events (participants affected / at risk) | 67/82 | 52/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours (N=82) | Medroxyprogesterone Acetate (MPA) (N=83)
Endometriosis (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levonorgestrel Intrauterine System (LNG IUS) 20µg Per 24 Hours (N=82) | Medroxyprogesterone Acetate (MPA) (N=83)
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 3 | 5
Flatulence (Gastrointestinal disorders) | 2 | 0
Fatique (General disorders) | 4 | 2
Irritability (General disorders) | 2 | 0
Vaginitis bacterial (Infections and infestations) | 9 | 3
Urinary tract infection (Infections and infestations) | 6 | 3
Sinusitis (Infections and infestations) | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 1
Bronchitis (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 3
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 3
IUCD complication (Injury, poisoning and procedural complications) | 2 | 0
Intra-uterine contraceptive device expelled (Injury, poisoning and procedural complications) | 2 | 0
Weight increased (Investigations) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Headache (Nervous system disorders) | 13 | 9
Depression (Psychiatric disorders) | 2 | 1
Libido decreased (Psychiatric disorders) | 2 | 3
Ovarian cyst (Reproductive system and breast disorders) | 10 | 2
Breast tenderness (Reproductive system and breast disorders) | 4 | 3
Pelvis pain (Reproductive system and breast disorders) | 4 | 2
Breast cyst (Reproductive system and breast disorders) | 3 | 1
Menorrhagia (Reproductive system and breast disorders) | 3 | 1
Uterine spasm (Reproductive system and breast disorders) | 3 | 1
Breast pain (Reproductive system and breast disorders) | 2 | 0
Coital bleeding (Reproductive system and breast disorders) | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 3
Genital discharge (Reproductive system and breast disorders) | 2 | 0
Metrorrhagia (Reproductive system and breast disorders) | 2 | 0
Vaginal discharge (Reproductive system and breast disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 5 | 5
Hypertension (Vascular disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator shall provide Sponsor an advanced copy of any proposed publication at least 60 days prior to the planned date of publication. Sponsor shall have 30 days to recommend changes. Institution and Principal Investigator agree that adoption of recommended changes shall not be unreasonably refused.